CLINICAL TRIAL: NCT05105009
Title: Furosemide and Creatinine Tubular Stress Test in Order to Measure Proximal Tubule Residual Function: is It Better Than GFR?
Brief Title: Furosemide and Creatinine Tubular Stress Test in Order to Measure Proximal Tubule Residual Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, Head of Nephrology, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-1131
Record Dates: First submitted 2020-03-11; First posted 2021-11-03 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Furosemide; Creatinine; Iohexol

STUDY DESIGN:
Intervention Model Description: all KDIGO stages and healthy volunteers (Kidney donors)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All KDIGO stages and healthy volunteers (Experimental): 15 healthy volunteers and 35 through all KDIGO stages.
  Interventions: Drug: Furosemide Injection; Drug: Creatinine Powder; Drug: Iohexol

INTERVENTIONS:
Drug: Furosemide Injection — * Furosemide Stress Test ( 1mg/kg in non diuretic users and 1.5 mg/kg in diuretic users).
  * Oral creatinine load using 5 grams of creatinine
  Other Names: Furosemide
Drug: Creatinine Powder — 5g of creatinine (Sigma) in 250 ml of water was taken orally
  Other Names: Creatinine
Drug: Iohexol — 5 ml iohexol (Omnipaque) intravenously

SUMMARY:
This is a two phase study. The first part will take place at the National Institute of Cardiology in Mexico, the second phase will be made in collaboration with the University of California San Diego and University of Minnesota.

This is a non blind experimental study, 72 patients with different stages of CKD from the outpatient unit of the institute will be included. Each patient will receive a furosemide stress test of 1 mg/kg in non diuretic users and 1.5 mg/kg in diuretic users, in addition of 5 grams of creatinine oral intake, as well as Iohexol 5ml IV to measure GFR. After the intervention, blood and urine samples will be drawn at baseline, 60 minutes, 180 minutes, and 240 min. Urine output will be maintained during the study by the intravenous administration of Hartman's solution 1 -2 ml/kg body weight every hour, in addition to the volume of urine output in the preceding hour plus oral water ingestion as tolerated.

Blood and urine will be analized to measure creatinine (blood and urine), then samples will be processed for measurement of furosemide (HPLC-Uv vis), indoxyl sulphate, p-cresol, hippurate, and iohexol (mass spectometry).

The aim of this stiudy is to asses the differences between GFR and proximal tubule function.

DETAILED DESCRIPTION:
Residual kidney function (RKF) its a critical tool in the CKD evolution and prognosis. It's well known that preserving RKF increases survival in patients with CKD.

Traditionally Glomerular Filtration Rate (GFR), and proteinuria have been the variables used to asses RKF, wich are glomerular residual function (GRF) variables. This glomerulocentric assestment of RKF has been challenged recently. It is knows that urea is not the principal uremic toxine, the protein boud uremic toxins are particullary important because it's elimination depends of the proximal tubular organic anionic transporters (OAT), and the organic cationic transporters (OCT). The functional integrity of this transporters are lost in advanced CKD stages, and it´s accumulation increases cardiovascular and renal damage because they activate proinflammatory citokines, increasing mortality, this was shown specially with the accumulation and clearance of hippurate and p-cresol independently of GFR.

The purpose of this study is to asses the functional capacity of two AOT (hOAT1, and hOAT3, that can be blocked by furosemide), and one OCT (OCT2 blocked by creatinine) using an stress test. The stress test will be performed in healthy subjects as well as in CKD from different stages. Protein bound uremic toxins such as indoxyl sulphate, p-cresol, and hippurate will be measured.

In the stress the typical furosemide stress test described previously by Mehta will be implemented, in addition to an oral load of 5 grams of creatinine oral load. This levels should be efficient enough to assess the functionality of the OCT2. A comparison between the tubular creatinine secretine to filtrated creatinine measuring GFR using Iohexol will be performed.

In conclusion this is a pilot study aimed to establish a practical methodology for the assesment of proximal tubular function.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Patients with CKD that attends to the outpatient clinic.
* Residual uresis of 500 mL

Exclusion Criteria:

* Patients younger than 18 years old.
* Increase of Cr in a rate of 0.5 mg/dL, or loss of more than 30% of previous GFR.
* Patients with cardiorrenal syndrome type 1.
* Patients with dilated miocardiopathy.
* Volume overload or incomplete voiding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Tubular Residual Kidney Function | 1 year
  To assess the functionallity of the hOAT1 and 3, and hOCT2 by stress test using furosemide and creatinine loads.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chávez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bullen AL, Fregoso A, Ascher SB, Shlipak MG, Ix JH, Rifkin DE. Markers of Kidney Tubule Dysfunction and Major Adverse Kidney Events. Nephron. 2023;147(12):713-716. doi: 10.1159/000531946. Epub 2023 Jul 31. PMID 37524063
- [Background] Liu BC, Tang TT, Lv LL, Lan HY. Renal tubule injury: a driving force toward chronic kidney disease. Kidney Int. 2018 Mar;93(3):568-579. doi: 10.1016/j.kint.2017.09.033. Epub 2018 Jan 17. PMID 29361307
- [Background] Armenta A, Madero M, Rodriguez-Iturbe B. Functional Reserve of the Kidney. Clin J Am Soc Nephrol. 2022 Mar;17(3):458-466. doi: 10.2215/CJN.11070821. Epub 2021 Nov 10. PMID 34759007
- [Background] Lowenstein J, Grantham JJ. Residual renal function: a paradigm shift. Kidney Int. 2017 Mar;91(3):561-565. doi: 10.1016/j.kint.2016.09.052. PMID 28202171
- [Background] Toth-Manikowski SM, Sirich TL, Meyer TW, Hostetter TH, Hwang S, Plummer NS, Hai X, Coresh J, Powe NR, Shafi T. Contribution of 'clinically negligible' residual kidney function to clearance of uremic solutes. Nephrol Dial Transplant. 2020 May 1;35(5):846-853. doi: 10.1093/ndt/gfz042. PMID 30879076
- [Background] Mair RD, Lee S, Plummer NS, Sirich TL, Meyer TW. Impaired Tubular Secretion of Organic Solutes in Advanced Chronic Kidney Disease. J Am Soc Nephrol. 2021 Nov;32(11):2877-2884. doi: 10.1681/ASN.2021030336. Epub 2021 Aug 18. PMID 34408065
- [Background] Koepsell H. Organic Cation Transporters in Health and Disease. Pharmacol Rev. 2020 Jan;72(1):253-319. doi: 10.1124/pr.118.015578. PMID 31852803
- [Background] Emami Riedmaier A, Nies AT, Schaeffeler E, Schwab M. Organic anion transporters and their implications in pharmacotherapy. Pharmacol Rev. 2012 Jul;64(3):421-49. doi: 10.1124/pr.111.004614. Epub 2012 Mar 28. PMID 22457399
- [Background] Rehberg PB. Studies on Kidney Function: The Rate of Filtration and Reabsorption in the Human Kidney. Biochem J. 1926;20(3):447-60. doi: 10.1042/bj0200447. No abstract available. PMID 16743679
- [Background] Rodriguez-Iturbe B, Herrera J, Marin C, Manalich R. Tubular stress test detects subclinical reduction in renal functioning mass. Kidney Int. 2001 Mar;59(3):1094-102. doi: 10.1046/j.1523-1755.2001.0590031094.x. PMID 11231365
- [Background] Shannon JA. THE RENAL EXCRETION OF CREATININE IN MAN. J Clin Invest. 1935 Jul;14(4):403-10. doi: 10.1172/JCI100691. No abstract available. PMID 16694314
- [Background] Koyner JL, Davison DL, Brasha-Mitchell E, Chalikonda DM, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Bennett MR, Kimmel PL, Seneff MG, Chawla LS. Furosemide Stress Test and Biomarkers for the Prediction of AKI Severity. J Am Soc Nephrol. 2015 Aug;26(8):2023-31. doi: 10.1681/ASN.2014060535. Epub 2015 Feb 5. PMID 25655065
- [Background] Rivero J, Rodriguez F, Soto V, Macedo E, Chawla LS, Mehta RL, Vaingankar S, Garimella PS, Garza C, Madero M. Furosemide stress test and interstitial fibrosis in kidney biopsies in chronic kidney disease. BMC Nephrol. 2020 Mar 6;21(1):87. doi: 10.1186/s12882-020-01721-z. PMID 32143585
- [Background] Wu W, Bush KT, Nigam SK. Key Role for the Organic Anion Transporters, OAT1 and OAT3, in the in vivo Handling of Uremic Toxins and Solutes. Sci Rep. 2017 Jul 10;7(1):4939. doi: 10.1038/s41598-017-04949-2. PMID 28694431
- [Background] Lim YJ, Sidor NA, Tonial NC, Che A, Urquhart BL. Uremic Toxins in the Progression of Chronic Kidney Disease and Cardiovascular Disease: Mechanisms and Therapeutic Targets. Toxins (Basel). 2021 Feb 13;13(2):142. doi: 10.3390/toxins13020142. PMID 33668632
- [Background] Eloot S, Schepers E, Barreto DV, Barreto FC, Liabeuf S, Van Biesen W, Verbeke F, Glorieux G, Choukroun G, Massy Z, Vanholder R. Estimated glomerular filtration rate is a poor predictor of concentration for a broad range of uremic toxins. Clin J Am Soc Nephrol. 2011 Jun;6(6):1266-73. doi: 10.2215/CJN.09981110. Epub 2011 May 26. PMID 21617084
- [Background] Tang J, Liu N, Zhuang S. Role of epidermal growth factor receptor in acute and chronic kidney injury. Kidney Int. 2013 May;83(5):804-10. doi: 10.1038/ki.2012.435. Epub 2013 Jan 16. PMID 23325080
- [Background] Sauvant C, Hesse D, Holzinger H, Evans KK, Dantzler WH, Gekle M. Action of EGF and PGE2 on basolateral organic anion uptake in rabbit proximal renal tubules and hOAT1 expressed in human kidney epithelial cells. Am J Physiol Renal Physiol. 2004 Apr;286(4):F774-83. doi: 10.1152/ajprenal.00326.2003. Epub 2003 Nov 25. PMID 14644751
- [Background] Caetano-Pinto P, Jamalpoor A, Ham J, Goumenou A, Mommersteeg M, Pijnenburg D, Ruijtenbeek R, Sanchez-Romero N, van Zelst B, Heil SG, Jansen J, Wilmer MJ, van Herpen CML, Masereeuw R. Cetuximab Prevents Methotrexate-Induced Cytotoxicity in Vitro through Epidermal Growth Factor Dependent Regulation of Renal Drug Transporters. Mol Pharm. 2017 Jun 5;14(6):2147-2157. doi: 10.1021/acs.molpharmaceut.7b00308. Epub 2017 May 24. PMID 28493713
- [Background] Hropot M, Fowler N, Karlmark B, Giebisch G. Tubular action of diuretics: distal effects on electrolyte transport and acidification. Kidney Int. 1985 Sep;28(3):477-89. doi: 10.1038/ki.1985.154. PMID 4068482
- [Background] Burki R, Mohebbi N, Bettoni C, Wang X, Serra AL, Wagner CA. Impaired expression of key molecules of ammoniagenesis underlies renal acidosis in a rat model of chronic kidney disease. Nephrol Dial Transplant. 2015 May;30(5):770-81. doi: 10.1093/ndt/gfu384. Epub 2014 Dec 18. PMID 25523450
- [Background] Bergwik J, Kristiansson A, Allhorn M, Gram M, Akerstrom B. Structure, Functions, and Physiological Roles of the Lipocalin alpha1-Microglobulin (A1M). Front Physiol. 2021 Mar 3;12:645650. doi: 10.3389/fphys.2021.645650. eCollection 2021. PMID 33746781
- [Background] Cheng CJ, Nizar JM, Dai DF, Huang CL. Transport activity regulates mitochondrial bioenergetics and biogenesis in renal tubules. FASEB J. 2024 May 31;38(10):e23703. doi: 10.1096/fj.202400358RR. PMID 38805156
- [Background] Karagiannidis AG, Theodorakopoulou MP, Pella E, Sarafidis PA, Ortiz A. Uromodulin biology. Nephrol Dial Transplant. 2024 Jun 28;39(7):1073-1087. doi: 10.1093/ndt/gfae008. PMID 38211973
- [Background] Horsch M, Beckers J, Fuchs H, Gailus-Durner V, Hrabe de Angelis M, Rathkolb B, Wolf E, Aigner B, Kemter E. Uromodulin retention in thick ascending limb of Henle's loop affects SCD1 in neighboring proximal tubule: renal transcriptome studies in mouse models of uromodulin-associated kidney disease. PLoS One. 2014 Nov 19;9(11):e113125. doi: 10.1371/journal.pone.0113125. eCollection 2014. PMID 25409434
- [Background] Schmit DJ, Carroll LJ, Eckfeldt JH, Seegmiller JC. Verification of separate measurement procedures where analytical determinations influence the clinical interpretation of GFR: Iohexol quantitation by HPLC and LC-MS/MS. Clin Biochem. 2019 May;67:16-23. doi: 10.1016/j.clinbiochem.2019.03.007. Epub 2019 Mar 21. PMID 30905584
- [Background] Seegmiller JC, Wolfe BJ, Albtoush N, Melena I, Gross SP, Vinovskis C, Ix JH, Bjornstad P. Tubular Secretion Markers, Glomerular Filtration Rate, Effective Renal Plasma Flow, and Filtration Fraction in Healthy Adolescents. Kidney Med. 2020 Aug 7;2(5):670-672. doi: 10.1016/j.xkme.2020.05.013. eCollection 2020 Sep-Oct. No abstract available. PMID 33089146
- [Derived] Madero M, Fernandez-Yepez AK, Resendiz-Albor AA, Rivera Chavez JA, Seegmiller JC, Rodriguez-Iturbe B. Estimation of Proximal Tubular Function by Stimulation of Organic Anion and Cation Transporters. J Am Soc Nephrol. 2025 Mar 24;36(9):1786-1797. doi: 10.1681/ASN.0000000686. PMID 40126554